CLINICAL TRIAL: NCT05987865
Title: EEG- or STN LFP-based Neurofeedback Training for Improving Motor Functions in Parkinson's Disease
Brief Title: Neurofeedback Training for PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: St George's London University Hospitals NHS Foundation Trust (Unknown); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 249990
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease; Healthy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People with Parkinson's disease or Healthy Control (Experimental): The experimental arm involves either patients with PD or healthy control, who will receive both experimental or non-experimental (control) intervention conditions.
  Interventions: Behavioral: Neurofeedback training

INTERVENTIONS:
Behavioral: Neurofeedback training — Features related to PD symptoms will be extracted from the brain recordings in real-time and used to drive a visual cursor on a computer screen placed in front of the participant, while the participant will be asked to try to control the cursor by regulating their brain signals.

SUMMARY:
The goal of this clinical trial is to test neurofeedback training in both people with Parkinson's disease and healthy control.

The main questions it aims to answer are:

* To demonstrate that EEG based or STN LFP based neurofeedback can help patients with Parkinson's disease to volitionally modulate pathological brain activities measured non-invasively;
* To evaluate the learning effect of the neurofeedback training with multiple training sessions

Patient participants will be asked to receive the research intervention called neurofeedback training for maximal three separate sessions. During the intervention, the participants will also be asked to press a pinch meter as fast as possible in order to measure the reaction time, meanwhile, different type of brain signals will be recorded.

. This will be a within-subject cross-over study contrasting the effect of the neurofeedback training and no training.

ELIGIBILITY:
Inclusion Criteria:

* Participants with symptomatic Parkinson's disease or age-matched healthy control
* Adequate understanding of verbal explanation or written information given in English
* Able and willing to give informed consent.
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Lack of capacity to consent (judged by the researcher taking consent as not having sufficient mental capacity to understand the study and its requirements)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
The feasibility of using EEG-based neurofeedback to help patients with Parkinson's disease to volitionally modulate pathological brain activities measured non-invasively. | 10 days
  The final position of the cursor and beta power changes after neurofeedback training will be measured and reported.
Learning effect of the neurofeedback training with multiple training sessions | 10 days
  The final positions of the cursor and the changes in beta power will be measured and compared across different training sessions.

SECONDARY OUTCOMES:
The effect of EEG-based neurofeedback on motor performance quantified as reaction time in patients with Parkinson's disease | 10 days
  The reaction time following cued motor task will be measured, and compared between training and no-training conditions.
The effect of EEG-based neurofeedback on motor performance quantified as peak movement velocity in patients with Parkinson's disease | 10 days
  The peak movement velocity during the cued motor task will be measured, and compared between training and no-training conditions.
The effect of EEG-based neurofeedback on parkinsonian tremor | 10 days
  The acceleration data will be measured from patient's arms during neurofeedback training, which will be used to quantity the tremor severity by looking at the power at patient specific tremor frequency band. The comparison on tremor severity between training and no-training conditions will be reported.
The effect of EEG-based neurofeedback on motor Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) score | 10 days
  MDS-UPDRS is a comprehensive 50 question assessment of both motor and non-motor symptoms associated with Parkinson's. Each question will be scored between 0 and 5, with a higher value indicates more severe assessment. In this study, the motor part of UPDRS scores on the patients will be measured, and compared before and after neurofeedback training.
The effect of EEG-based neurofeedback on motor performance quantified as reaction time in healthy age-matched control | 10 days
  The reaction time following cued motor task will be measured, and compared between training and no-training conditions in healthy age-matched control group.
The peak movement velocity during the cued motor task will be measured, and compared between training and no-training conditions in healthy age-matched control group. | 10 days
  This will be assessed by comparing the peak movement velocity during the cued motor task between training and no-training conditions.

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will share the fully anonymized brain recordings and behavioural data on the Oxford Research Archives or the MRC Brain Network Dynamics Unit Data Sharing platform.